CLINICAL TRIAL: NCT07210710
Title: CKD Awareness, Referrals, Education, and Support Intervention for Early-Stage CKD
Acronym: CARES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-0858; P30DK092949 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease; Diabetes
Keywords: chronic kidney disease; diabetes; chronic disease self-management; disease awareness; intervention; social determinants of health; motivation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — Referral and Consultation; Educational Status; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will participate in a nurse-led virtual session delivering education about chronic kidney disease, motivational interviewing to set a self-management goal, and screening/referral for social determinants of health barriers to treatment adherence and engagement.
  Interventions: Behavioral: CKD Awareness, Referrals, Education, and Support (CARES)
- Control group (Active Comparator): The attention control group will participate in a nurse-led virtual session delivering general information about diabetes and treatment.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: CKD Awareness, Referrals, Education, and Support (CARES) — We will target diabetic patients eligible for an early-stage CKD diagnosis with a nurse-delivered, pre-PCP-visit 1:1 virtual session including 1) tailored, evidence-based CKD education 2) motivational interviewing with self-management goal setting, and 3) social determinants of health screening with referrals to services as needed.
  Arms: Intervention group
Behavioral: Attention control — The control group will receive an attention control session of general education about diabetes-related health behaviors (e.g., diet and physical activity) that does not refer to CKD, based on American Diabetes Association materials.
  Arms: Control group

SUMMARY:
The goal of this pilot clinical trial is to learn if an intervention delivering education, motivational support, and social support can prevent worsening kidney disease in adults with diabetes and early-stage kidney disease. The main questions it aims to answer are:

1. Is this intervention feasible to deliver and acceptable to patients?
2. What is the impact of the intervention on patient motivation, self-efficacy, kidney disease knowledge, and use of support services referrals?

The investigators will compare information collected about participants' response to this intervention with a group of similar patients who receive general diabetes information.

Participants will meet virtually with a nurse approximately 1 week before a scheduled primary care provider visit and complete surveys over the phone three times in a period of three months.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) progression to kidney failure causes devastating declines in quality of life and mortality, with high healthcare costs. CKD affects ~15% of all adults in the U.S. and ~40% of adults with diabetes, with substantial variability in rate of progression to kidney failure. Negative social determinants of health (SDOH), such as food insecurity can speed up disease progression. However, if CKD progression to kidney failure can be prevented or delayed, patients can experience minimal impact on health and well-being. The diagnosis, treatment, and monitoring of early-stage, asymptomatic CKD occurs predominantly in the primary care setting, including for those with diabetes. Unfortunately, the rates of guideline-based CKD care delivery are low, and as a result, clinical diagnosis of early-stage CKD is as low as 50%. Delay in receiving a CKD diagnosis is associated with faster progression to kidney failure. Furthermore, because CKD is not always prioritized in the busy primary care setting, most patients are unaware they have CKD and have low rates of CKD knowledge, which impedes their ability to adhere to treatment. To address the issues of underdiagnosis, patients' lack of disease knowledge and self-efficacy, and the impact of SDOH for patients with diabetes and CKD, proactive action is critical. The investigators will target patients with diabetes who are eligible for an early-stage CKD diagnosis with a nurse-led, pre-primary care-visit 1:1 virtual session including evidence-based CKD education, motivational interviewing, and SDOH screening with referrals to services.

ELIGIBILITY:
Inclusion Criteria:

* adults (18+)
* diabetes diagnosis (type 1 or 2)
* CKD Stage 3 diagnosis eligible
* >1 prior visit at the UIHealth primary care clinics
* can speak English

Exclusion Criteria:

* CKD of congenital or pediatric onset
* history of kidney transplant
* cognitive impairment as documented in the medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Motivation for diabetes-related self-care behaviour scale | From enrollment to study completion (2-3 months)
  Participant self-report. A scale from 1-5, with a lower score meaning not motivated and a higher score meaning highly motivated. Items are different self-management behaviors (e.g., medication, diet, exercise).
Kidney Disease Knowledge Survey | From enrollment to study completion (2-3 months)
  Participant self-report. A set of fact-based questions about kidney disease which has a right and a wrong answer. Participants will be scored based on % correct answers.
CKD Self Efficacy Instrument | From enrollment to study completion (2-3 months)
  Participant self-report. The scale ranges from 1-10, with low scores indicating not at all confident and high scores indicating totally confident.
Social referral uptake | From enrollment to study completion (2-3 months)
  Participant self-report of uptake of any support services for barriers to treatment adherence that are needed.

SECONDARY OUTCOMES:
Brief Illness Perceptions Questionnaire | From enrollment to study completion (2-3 months)
  Participant self-report. Scale from 1-10, with the meaning of numbers changing per item. Assessing participants' perspective and understanding of their chronic condition. Items assessed individually or using clustering approaches.
Patient activation Measure | From enrollment to study completion (2-3 months)
  Participant self-report. Scales are 1-4 with a not applicable option, lower scores meaning less activated and engaged in care and higher scores meaning more activated and engaged in care.
PROMIS Medication Adherence Scale | From enrollment to study completion (2-3 months)
  Participant self-report. Scale from 1-5 indicating agree to disagree, with items about performance of medication adherence behaviors.
Dialysis Diet and Fluid Non-adherence Questionnaire | From enrollment to study completion (2-3 months)
  Participant self-report. One item asking how many days in the last week guidelines were not followed, and another item asking to what degree they were not followed, from completely to not at all.
International Physical Activity Questionnaire | From enrollment to study completion (2-3 months)
  Participant self-report. Scale is 1-7 indicating the number of days a type of physical activity was performed in the previous week. Items are different types of physical activity behaviors.
Care plan changes | From enrollment to study completion (2-3 months)
  review of EHR data related to PCP visit, assess if any CKD-related information or changes were documented
Protocol for Responding to and Assessing Patients' Assets, Risks, and Experiences | From enrollment to study completion (2-3 months)
  Participant self-report. Items and response options vary and ask questions about social determinants of health issues (e.g., food insecurity, housing insecurity). Screening tool with no scores.

IPD SHARING:
Plan to Share IPD: Yes
Data collected from participants includes: demographic, clinical history characteristics, comorbidity data, and new diagnoses or treatment plan changes will be collected through electronic medical record (EMR) abstraction. Social determinants of health barriers and uptake, self-efficacy, patient activation, motivation, treatment adherence, CKD knowledge, and CKD perceptions, feasibility, and acceptability quantitative data will be acquired through self-report questionnaires. All data will be collected in REDCap and de-identified prior to receipt by the repository, and a unique study identifier will be created for each subject.
  All deidentified quantitative study data that are not designated as restricted use by our repository, INtellectual property in DIGital form available online in an Open environment (INDIGO), will be shared openly.
Time Frame: All data will be shared the end of the award period or the time of an associated publication, whichever comes first. Publication-specific data will be shared when the pre-print is available. A DOI will aid in findability and the DOI will be included in relevant publications whenever possible. Study data deposited in INDIGO will be available to the research community in perpetuity.
Access Criteria: Users of the public use data must register with INDIGO and agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads.
URL: https://indigo.uic.edu/